CLINICAL TRIAL: NCT01421745
Title: Construct Validity, Responsiveness, and Demographic Predictors of the Inventory for Assessing the Process of Cultural Competence Among Healthcare Professionals - Student Version (IAPCC-SV)
Brief Title: Construct Validity, Responsiveness, and Demographic Predictors of the IAPCC-SV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Texas State University, San Marcos (Other); Texas Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Suzanna Dougherty Okere, Doctoral Candidate, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 16206
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Cultural Competence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cultural Competence Module (Experimental): The module will include lecture, case studies, and discussion of cultural competence.
  Interventions: Other: Cultural Competence Education module

INTERVENTIONS:
Other: Cultural Competence Education module — A four hour cultural competence education module including lecture, case studies, and discussion of cultural competence.

SUMMARY:
There are three purposes for this study:

I. to establish the construct validity (via factor analysis) of the Inventory for Assessing the Process of Cultural Competence Among Healthcare Professionals - Student Version (IAPCC-SV) II. to determine the responsiveness of the IAPCC-SV III. to investigate demographic predictor variables of the IAPCC-SV

It is hypothesized that:

I. the variables will load on only one component, with each component being represented by a number of strongly loaded variables II. the IAPCC-SV will demonstrate responsiveness, evidenced by significantly higher post-module IAPCC-SV scores of the experimental group when compared to the control group III. the cultural composite score and race will be significant predictors of IAPCC-SV score

ELIGIBILITY:
Inclusion Criteria:

* First semester PT students at Texas State will be eligible to participate in the study

Exclusion Criteria:

* Students previously enrolled in a PT education program will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Inventory for Assessing the Process of Cultural Competence Among Healthcare Professionals - Student Version (IAPCC-SV) Score | pre and post module

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna D Okere, MPT, Principal Investigator — Texas Woman's University
Locations (1):
- Texas State University-San Marcos, San Marcos, Texas, United States